CLINICAL TRIAL: NCT04371276
Title: Evaluation of the Seroepidemiology of Hepatitis A and B in the General Population for Informing the Development of New Hepatitis Vaccination Strategies in Hong Kong
Brief Title: Seroepidemiology of Viral Hepatitis in Hong Kong
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Shui-Shan Lee, MD, Professor, Chinese University of Hong Kong
Other Study IDs: 17160962
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Viral Hepatitis
Keywords: hepatitis A; hepatitis B; epidemiology
MeSH Terms: conditions — Hepatitis A; Hepatitis B | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — Blood samples will be collected from recruited subjects from invited households for testing for hepatitis B (HBsAg, anti-HBs and anti-HBc) and hepatitis A (anti-HAV)
  Other Names: blood sampling for serology testing

SUMMARY:
Immunisation policies have strong influences on the epidemiology of hepatitis A and B infection. In Hong Kong, vaccines against both viruses have been available through different channels and programmes in the past 3 decades. To evaluate the changes in the prevalence of hepatitis A and B in the general population, a seroepidemiology study is conducted involving a prospective cross-sectional survey followed for serology testing. Eligible members of 1327 spatially random households would be invited to join the study by completing a questionnaire and providing blood samples, either by dried blood spots or venesection, for determining the presence of antigen and/or antibody against hepatitis B, as well as antibody against hepatitis A. The main measures comprise a set of metrics on the prevalence of hepatitis A and B. Analysis would be conducted to examine the association of risk factors with the tested markers and describe the attitudes towards viral hepatitis vaccination. The results would allow us to understand the transmission potential of hepatitis A and B in the community would be influenced by the changing disease epidemiology and coverage of vaccination, which inform the development of new vaccination strategies in Hong Kong

ELIGIBILITY:
Inclusion Criteria:

* residents normally living in Hong Kong
* living in domestic households randomly selected from Building Groups
* Any age, while subjects below the age of 18 would require informed consent of their guardians for participation
* Any gender

Exclusion Criteria:

* unable to understand written Chinese or English,
* failure to give consent for participation
* living in institution or non-domestic housing,
* foreign domestic helpers,
* normally living in Hong Kong

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Residents of Building Groups from diverse geographical locations in Hong Kong selected through cluster sampling are targeted. With the building information available, three households would be randomly selected from each Building Group.
Sampling Method: Probability Sample
Enrollment: 2888 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
hepatitis B infection prevalence | 12 months
  Proportion of individuals with positive HBsAg
hepatitis A immunity prevalence | 12 months
  Proportion of individuals with positive IgG against HAV

CONTACTS AND LOCATIONS:
Overall Officials: Shui Shan Lee, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Poon CM, Chan DP, Lee SS, Wong NS. Seroepidemiology of hepatitis A and B in the general population in Hong Kong: protocol of a cross-sectional survey using spatial sampling in a highly urbanised city. BMJ Open. 2021 Mar 22;11(3):e042065. doi: 10.1136/bmjopen-2020-042065. PMID 33753433